CLINICAL TRIAL: NCT05295485
Title: Evaluation of the Course Format "NASIM25" - Development of Skills and Professional Safety of Aspiring Prehospital Emergency Physicians by the Course NASIM25
Brief Title: Evaluation of the Course Format "NASIM25"
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Thomas Ott, Thomas Ott, M.D., Principal Investigator, Department of Anesthesiology, University Hospital Center, Johannes Gutenberg University Mainz
Other Study IDs: 22-00708
Record Dates: First submitted 2022-03-06; First posted 2022-03-25 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Emergencies; Trauma Injury
Keywords: emergencies; trauma; pediatric emergencies; prehospital emergencies
MeSH Terms: conditions — Emergencies; Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators intend to evauate the development and professional safety of aspiring prehospital emergency pyhsicians in a cross sectional and longitudinal modality. This compass objecitve and subjective evaluable professional skills essential in prehospital emergency medicine.

DETAILED DESCRIPTION:
In the course format "NASIM25" aspiring prehospital emergency physicians are trained in 25 simulation based scenarios dealing about situations being rare on the scene having have a tremendous impact on the patients if not treated adequately.

To evaluate the impact of the course format on the skills of the participants (i.e. aspiring prehospital emergency physicians) the investigators quantify the trained skills and professional safety in three dimensions of skills and professional safety:

1. The influence on applying the ABCDE-Approach using the a validated score by Peran et al 2020 (ABCDE cognitive aid tool in patient assessment -development and validation in a multicenter pilot simulation study. BMC Emerg Med. 2020;20(1)) and non technical skills using a validated score by Kim et al 2009 (Kim J, Neilipovitz D, Cardinal P, Chiu M.A comparison of global rating scale and checklist scores in the validation of an evaluation tool to assess performance in the resuscitation of critically ill patients during simulated emergencies (abbreviated as "CRM simulator study IB"). Simul Healthc. 2009;4(1):6-16)
2. The influence on the cource on the self- and external assessement of the participants using school marks
3. The influence on the professional safety using a web based survey in a longitudinal modality throughout the entire qualification curriculum of prehospital emergency medicine.

ELIGIBILITY:
Inclusion Criteria:

* physician aspiring the qualification: "prehospital emergency physician" and participating in the course: NASIM25

Exclusion Criteria:

* not participating in the course NASIM25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: physicians that are aspiring the qualification: "prehospital emergency physician"
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Influence on applying the ABCDE-Approach and non-technical skills | 3 Days
  The investigators use a 33 item compassing checklist to quantify the ABCDE approach according to Peran et al. 2020 (Peran et al. ABCDE cognitive aid tool in patient assessment - development and validation in a multicenter pilot simulation study. BMC Emerg Med. 2020;20(1):95.) and a 7 items compassing Ottawa Global scale to quantify the non-technical skills concerning CRM according to Kim et al. 2009 (Kim et al. A comparison of global rating scale and checklist scores in the validation of an evaluation tool to assess performance in the resuscitation of critically ill patients during simulat-ed emergencies (abbreviated as "CRM simulator study IB"). Simul Healthc. 2009;4(1):6-16.). Further details are cited in the study description -> Detailed description
Influence on self- and external assessement | 3 Days
  The investigators use school marks (1=best, 6=worst) to quantify the global performance of the participants to rate the performance at the end of each scenario within the course for external assessment and the same school marks as an internal self-assessment given by the participants.
  Further details are cited in the study description -> Detailed description
Influence on the professional safety | 1 Year
  The investigators use a self-designed questionnair compassing 25 diseases. Every participant has to self-assess the own capability to handle each of the diseases in a 10 items likert scale (1: very unsafe in handling, 10: very safe in handling) over the points in time: before the course, after the course and after an additional time frame after the course.

CONTACTS AND LOCATIONS:
Overall Officials: Ott Thomas, M.D., Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- University Hospital Centre Mainz, Mainz, RLP, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peran D, Kodet J, Pekara J, Mala L, Truhlar A, Cmorej PC, Lauridsen KG, Sari F, Sykora R. ABCDE cognitive aid tool in patient assessment - development and validation in a multicenter pilot simulation study. BMC Emerg Med. 2020 Dec 4;20(1):95. doi: 10.1186/s12873-020-00390-3. PMID 33276731
- [Result] Kim J, Neilipovitz D, Cardinal P, Chiu M. A comparison of global rating scale and checklist scores in the validation of an evaluation tool to assess performance in the resuscitation of critically ill patients during simulated emergencies (abbreviated as "CRM simulator study IB"). Simul Healthc. 2009 Spring;4(1):6-16. doi: 10.1097/SIH.0b013e3181880472. PMID 19212245
- See also: official website providing informations about the course NASIM25 — https://www.unimedizin-mainz.de/anaesthesiologie/klinische-partner/simulationszentrum/nasim25.html